CLINICAL TRIAL: NCT00213265
Title: Safety and Immunogenicity of 7-Valent Pneumococcal Conjugate Vaccine Among Solid Organ Transplant Recipients: Protocol 1A and 1B
Brief Title: Safety and Immunogenicity of 7-Valent Pneumococcal Conjugate Vaccine in Children Receiving Solid Organ Transplants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Upton Allen, Chief, Division of Infectious Diseases, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0020020011
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Organ Transplant; Immunosuppression
Keywords: organ transplantation; immunosuppression; vaccine; pneumococcal conjugate vaccine; pediatrics
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Biological: Pneumococcal 7-valent Conjugate Vaccine
- 2 (Experimental)
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 7-valent pneumococcal conjugate vaccine — For transplant patients, vaccination will be started at 4 months or greater after transplantation. The second dose will be given 8 weks following the frist, the third dose 8 weeks after the second, and the fourth will be given 8 weeks after the third.
  Other Names: Prevnar
  Arms: 2
Biological: Pneumococcal 7-valent Conjugate Vaccine — Healthy infants: The Prevnar schedule for healthy infants consists of 3 doses of 0.5 ml each, at approximately 2 month intervals, followed by a fourth dose of 0.5 ml at 12-15 months of age (i.e., 2, 4, 6, and 12-15 months)
  Previously unvaccinated older infants and children, who are beyond the age of the routine infant schedule, should receive the follwong schedule:
  7-11 months of age: 3 doses (2 doses at least 4 weeks apart with the third dose after the first birthday and separated from the second dose by at least two months)
  12-23 months of age: 2 doses (at least 2 months apart)
  ≥24 months through 9 years of age: 1 dose
  Other Names: Prevnar
  Arms: 1

SUMMARY:
We plan to study whether the 7-valent pneumococcal conjugate vaccine (Prevnar™) is safe and effective in protecting children who have had a solid organ transplantation and healthy children from pneumococcal infections.

We expect that two or more doses of Prevnar™ will result in similar antibody responses among transplant recipients compared with healthy control subjects, and that children who have undergone solid organ transplant will have a similar number of serious vaccine-related adverse events within 7 days after Prevnar™ as the healthy patients.

DETAILED DESCRIPTION:
Solid organ transplantation (SOT) has emerged as a lifesaving therapy for many patients with end organ failure. SOT recipients have a lifelong increased risk for infections as a result of immunosuppression, including those caused by pneumococci. The increased susceptibility to pneumococcal infections is multi-factorial and is related to underlying immunosuppression as well as varying degrees of splenic dysfunction as a result of underlying pretransplantation diseases, among other factors.

The types and severity of invasive pneumococcal disease vary among each transplant population. However, comparative data are lacking. Lung transplant recipients have the highest incidence of bacterial pneumonia among solid organ transplant recipients. Pneumonia secondary to Streptococcus pneumoniae occurs in heart transplant patients at a rate 10 times that found in the general population. It is suggested that besides the intensity of immunosuppression, ongoing immunosuppression is important as a risk factor for invasive pneumococcal disease in transplant recipients.

Despite the fact that 23-valent polysaccharide pneumococcal vaccine is one of the vaccines that receives priority among organ transplant recipients, at the Hospital for Sick Children, several cases of pneumococcal disease have been seen. The advent of the 7-valent conjugate vaccine affords the opportunity to possibly reduce the burden of pneumococcal disease in the patient population by virtue that it may be more immunogenic in transplant patients

This study will examine the antibody titres achieved among transplant recipients who are immunized with Prevnar™, as well as evaluate the safety and tolerability or Prevnar™ administered as a three-dose regimen to children and adolescents following organ transplantation.

ELIGIBILITY:
Inclusion Criteria:

Transplant recipients:

* Children 4 months of age up to 18 years of age
* received a kidney, liver, heart, lung or other solid organ transplantation in a Canadian transplant centre
* Informed consent obtained

Healthy Infants and Children:

* Children 2 months to 9 years of age
* no underlying chronic medical conditions
* Informed consent obtained

Exclusion Criteria:

* Previous immunization with pneumococcal vaccine.
* Known hypersensitivity to any of the components of the vaccine, including diphtheria toxoid. Besides the saccharides and CRM197 carrier protein, the vaccine contains aluminum phosphate adjuvant.
* Any significant infection and/or fever at the time of vaccination
* Major acute illness such as clinical instability and acute graft rejection
* Latex allergy

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2002-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Concentration of pneumococcal antibodies | Transplant patients: at baseline, just before dose 3, and 6-8 weeks after dose 3; Controls: at baseline, just before dose 3, and 6-8 weeks after dose 3. For those whose series consisted of 1 or 2 doses, at baseline, and 6-8 weeks after doses 1 and 2.
Serious vaccine related adverse events | 7 days post-vaccination

SECONDARY OUTCOMES:
Nature of immune suppression | 24-28 weeks
Presence of bacterial, viral or other opportunistic infections | 24-28 weeks
Presence of rejection after enrollment | 24-28 weeks
Presence of concurrent diseases or conditions including alterations of renal, hepatic, cardiac and bowel function | 24-28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Upton Allen, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada; Upton Allen, Study Chair — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada